CLINICAL TRIAL: NCT06463561
Title: Effect of 12 Months of Treatment With Continuous Positive Airway Pressure on Lipid Profile and Hyperuricemia in Patients With Dyslipidemia and Moderate-severe Obstructive Sleep Apnea. A Randomized, Open-labell, Parallel Clinical Trial
Brief Title: CPAP Effect on Lipid Profile and Hyperuricemia in Patients With Dyslipidemia and Moderate-severe Obstructive Sleep Apnea
Acronym: CPAPLIP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario del Henares (Unknown)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, PhD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 082024
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-06

CONDITIONS: Sleep Apnea; Dyslipidemias; Hyperuricemia
MeSH Terms: conditions — Sleep Apnea Syndromes; Dyslipidemias; Hyperuricemia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Conventional hygienic-dietary recommendations and promotion of daily physical activity
  Interventions: Other: Hygienic-dietary recommendations and daily physical activity promotion
- CPAP group (Experimental): Conventional hygienic-dietary recommendations and promotion of daily physical activity, plus treatment with positive airway pressure (CPAP)
  Interventions: Device: Continuous positive airway pressure; Other: Hygienic-dietary recommendations and daily physical activity promotion

INTERVENTIONS:
Device: Continuous positive airway pressure — Treatment will start with an empirical pressure of 8 cmH2O and, within a maximum of 3 weeks, the pressure will be adjusted by means of automatic titration, establishing the pressure corresponding to the 95th percentile.
  Arms: CPAP group
Other: Hygienic-dietary recommendations and daily physical activity promotion — Hygienic-dietary recommendations on sleep and intervention for the promotion of daily physical activity, establishing walking as a goal 10,000 steps per day. To do this, they will be provided with a pedometer and asked to fill out a form with the steps walked each day. At each visit, the distance walked will be reviewed and the goal set will be reiterated.

SUMMARY:
Clinical Trial Phase IV Indication: Moderate-severe obstructive sleep apnea and dyslipidemia.

Objectives:

Main objective: To test whether 12 months of CPAP treatment associated with conventional pharmacological treatment improves the lipid profile of patients with dyslipidemia and moderate to severe OSA.

Secondary objectives:

* To test whether 12 months of treatment with CPAP associated with conventional pharmacological treatment improves serum uric acid concentration in patients with dyslipidemia and moderate-severe OSA.
* To determine the additional medium- and long-term effect of CPAP on insulin resistance in patients with dyslipidemia and moderate-severe OSA.
* To evaluate the impact of CPAP treatment on cardiovascular risk reduction in patients with dyslipidemia and moderate-severe OSA.
* To analyze the impact of supplemental CPAP treatment on glycemic control and C-reactive protein concentration in patients with dyslipidemia and moderate-severe OSA.
* To establish the impact of supplemental CPAP therapy on health-related quality of life in patients with dyslipidemia and moderate-severe OSA.
* To evaluate the effect of CPAP on inflammatory cytokines, oxidative stress biomarkers, sympathetic tone and intake-regulating hormones in patients with dyslipidemia and moderate-severe OSA.
* To relate CPAP-induced changes in serum lipid and uric acid concentration to changes in basal inflammatory response, oxidative stress, sympathetic activity, and intake-regulating hormones.
* To identify the subgroup of patients with dyslipidemia and moderate-severe OSA in whom 12 months of CPAP treatment achieves a more marked reduction in serum lipids and uric acid.

Design Randomized, parallel-group, nonblinded, controlled clinical trial with conventional treatment.

Study population Subjects aged 35 to 80 years with a diagnosis of dyslipidemia made at least six months ago and with moderate-severe obstructive sleep apnea (OSA) not requiring CPAP treatment according to conventional indications.

Sample size: 110 patients in each treatment arm.

Treatment Patients will be randomly assigned in a 1:1 ratio to one of the following treatment arms:

1. Conventional hygienic-dietary recommendations and promotion of daily physical activity.
2. Conventional hygienic-dietary recommendations and promotion of daily physical activity, plus treatment with positive airway pressure (CPAP).

Efficiency variables

* Main variables: LDL-cholesterol and uric acid.
* Total cholesterol, HDL-cholesterol and triglycerides.
* Basal blood glucose, glycosylated hemoglobin (HbA1c), creatinine and C-reactive protein.
* Systemic biomarkers: inflammatory (IL-6, IL-8 and TNF-α), oxidative stress (8-isoprostane), endothelial damage (endothelin, VCAM-1 and ICAM-1), sympathetic activity (neuropeptide Y) and appetite-regulating hormones (leptin, orexin A/hypocretin 1 and ghrelin).
* Clinical questionnaires: SF-12, EuroQoL, FOSQ and IPAQ.

Safety variables

* Clinical adverse event reporting.
* CPAP compliance (average hours of use per day).
* Epworth Sleepiness Questionnaire.
* Development of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 35 to 80 years old
* Diagnosis of dyslipidemia. It will be considered as such, the existence of a previous clinical record of a diagnosis of dyslipidemia associated with treatment with lipidlowering agents, treatment with lipid-lowering agents or the presence of an altered blood test in the last two months, using the following cut-off points: total cholesterol ≥ 200 mg/dl, triglycerides ≥ 180 mg/dl, HDL-cholesterol ≤ 40 mg/dl or LDL-cholesterol ≥ 150 mg/dl.
* Moderate-severe sleep apnea, defined by AHI > 15 h-1 .

Exclusion Criteria:

* Predominance of central apneas-hypopneas, defined as more than 25% of total respiratory events.
* Patients with indications for CPAP treatment according to the International Sleep Consensus: hypertensive, excessive daytime sleepiness (Epworth Sleepiness Scale > 11) or impaired sleep-related quality of life considered relevant by their regular physician.
* Professional drivers, at-risk profession or respiratory insufficiency (according to criteria of the clinical pathway for the diagnosis and treatment of sleep-disordered breathing).
* Pretreatment with CPAP

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
CPAP effect on lipid profile | 12 months
  Comparison of 12-months change from baseline in the plasma level of LDL-cholesterol between the two study groups
CPAP effect on lipid profile-2 | 12 months
  Comparison of 12-months change from baseline in the plasma level of HDL-cholesterol between the two study groups
CPAP effect on lipid profile-3 | 12 months
  Comparison of 12-months change from baseline in the plasma level of total cholesterol between the two study groups
CPAP effect on lipid profile-4 | 12 months
  Comparison of 12-months change from baseline in the plasma level of triglycerides between the two study groups

SECONDARY OUTCOMES:
CPAP effect on uric acid | 12 months
  Comparison of 12-months change from baseline in the plasma level of uric acid between the two study groups
Medium-term CPAP effect on insulin resistance | 6 months
  Comparison of 6-months change from baseline in the HOMA index between the two study groups
Long-term CPAP effect on insulin resistance | 12 months
  Comparison of 12-months change from baseline in the HOMA index between the two study groups
CPAP effect on cardiovascular risk | 12 months
  Comparison of 12-months change from baseline in the cardiovascular risk score between the two study groups
CPAP effect on glycemic control | 12 months
  Comparison of 12-months change from baseline in the plasma level of HbA1c between the two study groups
CPAP effect on C-reactive protein | 12 months
  Comparison of 12-months change from baseline in the plasma level of C-reactive protein between the two study groups
CPAP effect on sleepiness | 12 months
  Comparison of 12-months change from baseline in the Epworth sleepiness scale between the two study groups
CPAP effect on health-related quality of life | 12 months
  Comparison of 12-months change from baseline in the EuroQoL score between the two study groups
CPAP effect on health-related quality of life-2 | 12 months
  Comparison of 12-months change from baseline in the SF-12 score between the two study groups
CPAP effect on daily physical activity | 12 months
  Comparison of 12-months change from baseline in the iPAQ score between the two study groups
CPAP effect on inflammatory cytokines | 12 months
  Comparison of 12-months change from baseline in the plasma levels of IL-6, IL-8 and TNF-α between the two study groups
CPAP effect on oxidative stress biomarkers | 12 months
  Comparison of 12-months change from baseline in the plasma level of 8-isoprostane between the two study groups
CPAP effect on sympathetic tone | 12 months
  Comparison of 12-months change from baseline in the plasma level of neuropeptide Y between the two study groups
CPAP effect on intake-regulating hormones | 12 months
  Comparison of 12-months change from baseline in the plasma levels of leptin, orexin A/hypocretin 1 and ghrelin between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Maria Angeles Ruiz-Cobos, MD, Study Chair — Hospital Universitario del Henares; Ana De la Rocha Prieto, MD, Principal Investigator — Hospital Universitario del Henares; Julia Dorta Díez de la Lastra, MD, Principal Investigator — Hospital Universitario del Henares; Raquel Casitas, MD, Principal Investigator — Hospital Universitario La Paz; Marina Blanco Cruz, ND, Principal Investigator — Hospital Universitario del Henares
Locations (1):
- Hospital Universitario del Henares, Coslada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided